CLINICAL TRIAL: NCT01865955
Title: Comparison Between Palpatory and Preprocedural Ultrasound Guided Techniques on Performance of Spinal Anesthesia in Term Parturients Undergoing Elective Caesarian Section- A Randomized Control Trial
Brief Title: Comparison Between Palpatory and Preprocedural Ultrasound Guided Techniques on Performance of Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-02
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Pregnancy
Keywords: Ultrasound; Spinal anesthesia; Cesarean section
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palpation (No Intervention): Palpation will be used to determine placement of the spinal needle.
- Ultrasound (Experimental): Ultrasound will be used prior to placement of the spinal needle.
  Interventions: Procedure: Ultrasound; Device: The spinal needle

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound applied to the lumbar region to determine spinal needle placement.
  Arms: Ultrasound
Device: The spinal needle
  Arms: Ultrasound

SUMMARY:
Pre-procedural ultrasound for Spinal & Epidural anesthesia is now being increasingly performed worldwide. Pre-procedural ultrasound assessment of the spine has been shown to facilitate the placement of epidural anesthesia in pregnant women, diagnostic lumbar punctures, performance of spinal anesthesia in non-obstetric patients and accurate identification of the interspace at which the puncture is being performed. This is especially important during spinal anesthesia, where puncture below the ending of the spinal cord is recommended for safety.

The purpose of this study is to compare the performance of spinal anesthesia between the pre-procedural ultrasound assessment of the spine and the traditional palpatory technique, in term pregnant women undergoing elective cesarean delivery. Furthermore, we aim to describe sonoanatomic features of the spine that could predict the ease of insertion of spinal anesthesia in that patient population.

We hypothesize that in term pregnant women undergoing elective cesarean delivery, pre-procedural ultrasound assessment of the spine will improve the success rate of spinal anesthesia at first attempt, compared to the traditional palpatory technique.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients scheduled to receive spinal anesthesia for elective cesarean sections
* ASA physical status 1 - 3
* Written informed consent
* Gestational age ≥ 37 weeks.

Exclusion Criteria:

* Patient's refusal.
* Body mass index ≥ 45
* Patient with marked spinal bony deformity (Severe scoliosis on visual inspection and previous spinal instrumentation).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Spinal needle redirections | 15 minutes
  Number of redirections needed to perform a successful spinal puncture (presence of cerebrospinal fluid). A needle redirection is defined as any change in needle insertion trajectory that did not involve complete withdrawal of the needle from the patient's skin. The first needle pass will not be considered a redirection.

SECONDARY OUTCOMES:
Needle reinsertions | 15 minutes
  Number of needle reinsertions defined as complete withdrawal of the spinal needle to the patient's skin followed by a new attempt in the same interspace.
Need to change to another interspace. | 15 minutes
  Relocating the spinal needle to another interspace.
Procedure time | 15 minutes
  Time taken to perform the spinal anesthesia, measured from insertion of the introducer needle to visualization of spinal fluid.
Pain score | 15 minutes
  Verbal Numerical Pain Scores during the procedure (0-10, where 0 means no pain and 10 mean the worst pain imaginable).
Intervertebral level agreement | 3 hours
  Intervertebral level agreement between L3-L4 obtained in the postoperative ultrasound assessment and the marked intervertebral level obtained pre-procedure, either by ultrasound or palpation.
Ultrasound Grading | 3 hours
  Ultrasound Grading: The image pattern of the intervertebral space will be categorized into three grades by three study investigators not involved in providing the spinal anesthesia: Typical Image,Atypical Image or Inconclusive Image.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Arzola, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada